CLINICAL TRIAL: NCT03390998
Title: Angiographic and Psychosocial Evaluation of Peripartum vs. Non Peripartum Spontaneous Coronary Artery Dissection (SCAD): A Collaborative Study
Brief Title: Angiographic and Psychosocial Evaluation of Peripartum vs. Non: SCAD
Acronym: SCAD
Status: Completed | Type: Observational
Sponsor: Katharine Sears Edwards (Other)
Collaborators: Massachusetts General Hospital (Other); Mayo Clinic (Other); University Hospital, Clermont-Ferrand (Other); University of British Columbia (Other); University of Leicester (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Katharine Sears Edwards, Clinical Assistant Professor, Medicine - Cardiovascular Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 40486
Record Dates: First submitted 2017-12-13; First posted 2018-01-05 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Spontaneous Coronary Artery Dissection
Keywords: Pregnancy-related SCAD; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peripartum SCAD: Female patients who experienced any SCAD event that occurred during pregnancy or up to 1 year post-delivery
- Non-peripartum SCAD: Female patients who experienced any SCAD with event onset outside of the pregnancy period

SUMMARY:
This multi-site international clinical research project is a collaboration between investigators from multiple institutions in the USA, Canada, and Europe. Approximately 7 to 11 sites will participate and provide data for analysis. Clinical operations (for data collection and analysis) across sites will be managed by Stanford. The study purpose is to determine differences in clinical and imaging presentation, in-hospital management and prognosis in peripartum and non-peripartum SCAD patients.

DETAILED DESCRIPTION:
There is a reason to believe that female sex hormone fluctuations during the peripartum period are linked with the occurrence of SCAD, and may be associated with a distinctive clinical presentation. In addition, symptoms of psychological distress may be linked to the development of SCAD and post-event distress is higher in SCAD patients than in those with coronary artery disease (CAD).

The primary objective is to determine differences in clinical and imaging presentation, in-hospital management and prognosis in peri-partum and non-peri-partum SCAD patients. At the methodological level, the purpose is to apply a systematic image analysis protocol for classifying SCAD lesions and to pool data to achieve adequate statistical power.

The secondary objective is to gather more information about psychological and psychosocial factors in SCAD patients. Specifically, to assess pre-event stress and psychological diagnoses and determine differences in post-event distress between peripartum and non-peripartum SCAD.

It is expected that these aims will result in two important outcomes. First, implementation of a systematic image analysis protocol for SCAD data will lead to improved reliability and, we expect, the detection of clinically meaningful differences between peripartum and non-peripartum SCAD. These differences may align with potential causal mechanisms for further study to ultimately better understand SCAD and develop treatment(s). Second, by characterizing the psychological distress experienced by SCAD patients, and differences between patients who experienced peripartum vs. non-peripartum SCAD, psychosocial risk factors may be identified and psychosocial interventions can be tailored to meet the needs of this unique patient population.

This is an observational study using cross-sectional design. There are two main components: a retrospective collection of medical history pertaining to SCAD event and prospective questionnaires. Sites may elect not to contact patients and not collect the prospective questionnaire.

Clinical variables will include demographic data, cardiac risk factors, medications and details of presentation (including peak troponin, left ventricular ejection fraction (LVEF), and days to discharge), as well as follow-up data, including recurrent events, and symptoms of depression, anxiety, stress, and PTSD.

Clinical data will be obtained by study collaborators and entered into a secure database maintained on Stanford systems. De-identified imaging data will be uploaded by collaborators. Imaging data will be analyzed by two independent readers (selected from participating institutions).

ELIGIBILITY:
Inclusion Criteria:

Sites contacting patients and/or conducting the survey

* Female adults 18 years of age and older
* Voluntary participation
* Patients with a known or suspected diagnosis of SCAD
* Ability to read in English
* Ability to access online consent and questionnaire portal

Sites not contacting patients and/or conducting the survey

* Female adults 18 years of age and older
* Patients with a known or suspected diagnosis of SCAD

Exclusion Criteria

- Not fulfilling inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women will be studied as the primary question relates to pregnancy-related SCAD
Study Population: Participants with pregnancy-related and non pregnancy-related SCAD will be recruited from the population of SCAD patients known to an international collaborative of investigators. We expect to enroll approximately 400 patients, 100 of whom have experienced peripartum SCAD. For each enrolled participant with peripartum SCAD, we will enroll 3 patients with non-peripartum SCAD who are the closest match on age at SCAD event and country.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
First Major Adverse Cardiovascular Event (post-SCAD) | First SCAD event represents t=0. Time (in days) from t=0 until the first occurrence of any of the above, for up to 6-months after t=0.
  The time from the first SCAD event until the first occurrence of (1) myocardial infarction, (2) re-vascularization, (3) stroke, or (4) death due to cardiovascular cause.

SECONDARY OUTCOMES:
Depression | At survey administration (post-SCAD), ranging from 6-months to 10 years post SCAD.
  Patient Health Questionnaire (PHQ9) is a 9-item questionnaire that measures depression on a scale of 0-27 (where >20 is major depression).
Anxiety | At survey administration (post-SCAD), ranging from 6-months to 10 years post SCAD.
  Generalized Anxiety Disorder (GAD-7) is a 7-item questionnaire that measures anxiety on a scale of 0-21 (where >14 is severe anxiety).
Stress | At survey administration (post-SCAD), ranging from 6-months to 10 years post SCAD.
  Perceived Stress Scale (PSS) is a 10-item questionnaire that measures stress on a scale of 0-40 (where >26 is high perceived stress).
Post-Traumatic Stress Disorder | At survey administration (post-SCAD), ranging from 6-months to 10 years post SCAD.
  PTSD CheckList (PCL-5) is a 20-item questionnaire that assesses the presence and severity of PTSD symptoms on a scale of 0-80 (where >32 suggests the patients needs further assessment to confirm a diagnosis of PTSD).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ann Tremmel, MD, MS, Principal Investigator — Stanford University; Katharine S. Edwards, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States